CLINICAL TRIAL: NCT02753959
Title: Changes in Regional Lung Ventilation Following Mechanical Insufflation-Exsufflation
Acronym: MIE and EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: B&D Electromedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PM Mar 16
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2018-04

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute Intervention (Experimental): Patients will need to be Clinically stable patients with established neuromuscular disease with clinical secretions or cough PEF <270 and history of chest infections. Patients are required to be stable for the preceding 4 weeks with no changes to medications or ventilator settings.
  Interventions: Other: Acute Intervention
- Stable Intervention (Experimental): Patients with established neuromuscular disease admitted to either the Lane Fox Respiratory Unit or Critical Care at St Thomas' Hospital with acute respiratory deteriorations and with the need for respiratory physiotherapy for secretion management.
  Interventions: Other: Stable Intervention

INTERVENTIONS:
Other: Acute Intervention — Patients will be set up onto their Non Invasive Ventilator and assessed for an hour prior to, during and following secretion clearance and will have the following assessed:
  * Electrical impedance tomography (EIT)
  * EMGpara
  * SpO2
  * tcCO2
  * Respiratory inductance plethysmography
  * EIT will be performed as 2 to 10-minutes recording of quiet breathing before and after each intervention
  Interventions will be set as follows with a 30 minute washout period between modes:
  * Manual techniques only
  * MIE at low pressure (+30 to -30)
  * MIE at high pressure (+60 to -60)
  Arms: Acute Intervention
Other: Stable Intervention — Patients will be set up onto their Non Invasive Ventilator and assessed for an hour prior to, during and following secretion clearance and will have the following assessed:
  * Electrical impedance tomography (EIT)
  * EMGpara
  * SpO2
  * tcCO2
  * Respiratory inductance plethysmography
  * EIT will be performed as 2 to 10-minutes recording of quiet breathing before and after each intervention
  Interventions will be set as follows with a 30 minute washout period between modes:
  * Manual techniques only
  * MIE at low pressure (+30 to -30)
  * MIE at high pressure (+60 to -60)
  Arms: Stable Intervention

SUMMARY:
Patients with NMD can suffer from a range of respiratory problems due to respiratory muscle weakness. Cough muscle weakness worsens secretion clearance from the airways, and increases the risk of infection. As a result, these patients often require chest physiotherapy or are supported with devices to aid clearance (such as mechanical insufflation-exsufflation) to reduce the risk of infection. Although evidence supports the use of these devices, the optimal technique or settings on the device are not clear.

Electrical impedance tomography (EIT) is a new technology that involves wearing a belt of sensors around the chest that provides information on how well the lungs are being filled with air. It allows a non-invasive assessment of the effect of each secretion clearance technique on lung ventilation in real-time.

This study aims to compare how well the lung is filled with air between three different techniques for secretion clearance (clearing mucus and phlegm from the airways), in order to determine which of the techniques is the most effective, in patients with NMD.

DETAILED DESCRIPTION:
Electrical Impedance Tomography (EIT) is a non-invasive, bedside monitoring technique that provides semi-continuous, real-time information about the regional distribution of the changes in electrical resistivity of the lung tissue due to variations in ventilation in relation to a reference state.

Information is gained by repeatedly injecting small alternating electric currents (usually 5 mA) at high frequency of 50 - 80 kHz through a system of skin electrodes (usually 16) applied circumferentially around the thorax in a single plane between the 4th and 6th intercostal space. While an adjacent pair of electrodes 'injects' the current ('adjacent drive configuration'), all the remaining adjacent passive electrode pairs measure the differences in electric potential. A resistivity (impedance) image is reconstructed from this data by a mathematical algorithm using a two dimensional model and a simplified shape to represent the thoracic cross-section.

The resulting image possesses a high temporal and functional resolution making it possible to monitor dynamic physiological phenomena (e.g., delay in regional inflation or recruitment) on a breath by breath basis. It is important to realize that the EIT images are based on image reconstruction techniques that require at least one measurement on a well-defined reference state. All quantitative data are related to this reference and can only indirectly quantify (relative) changes in local lung impedance (but not absolute).

Patients with respiratory muscle weakness have reduced cough strength and this can cause difficulties with clearing respiratory secretions. This impaired secretion clearance can lead to respiratory infections and acutely can causing small airway occlusion with subsequent ventilation-perfusion mismatch adversely effecting pulmonary mechanics. The use of cough assist devices, such as mechanical insufflation-exsufflation (MIE) can improve secretion clearance. Although there is evidence that these devices can improve secretion clearance the optimal pressures or technique required to provide effective secretion clearance is not known. Furthermore the use of high pressure swings that are now frequently used in clinical practice could lead to lung derecruitment. The use of EIT would allow a novel and effective method of assessing the ability to clear secretions and optimise ventilated lung in neuromuscular patients with poor cough and assess post procedure derecruitment.

MIE: A pilot physiological study will be performed in patients with neuromuscular disease with acute (10 patients) and chronic (10 patients) secretion management issues that require clinical use of MIE. These patients will be studied using 3 different clearance strategies low pressure MIE, higher pressure MIE and standard airway techniques. The project will assess differences in regional ventilation following augmented airway clearance and inform potential endpoints and feasibility for a larger trial regarding speed of recovery from respiratory infections in patients with neuromuscular disease.

There is a paucity of data regarding the physiological efficacy of MIE devices and although clinical consensus regards them as a beneficial adjunct to the management of patients with respiratory muscle weakness causing a reduction in effective secretion clearance it is less clear the optimum protocol to achieve secretion clearance. The aim of chest physiotherapy is to achieve clearance of airway secretions and allow improved gas exchange by enhancing ventilation and perfusion matching within the lung. The data suggesting optimum pressures for MIE are based around early work on achieving enhanced cough peak expiratory flow. More recently higher pressures have been suggested to achieve enhanced airway clearance. There may be potential beneficial effects with high pressure MIE by enhancing airway opening during the insufflation pressure achieving a degree of lung volume recruitment. Conversely, high insufflation pressures may adversely affect both pulmonary and cardiac physiology which may be further impacted by the large pressure swing during exsufflation. This is particularly relevant given the increasing co-morbid cardiomyopathy that occurs in many congenital neuromuscular diseases.

The initial phase of the project would be to generate pilot data with a comprehensive physiological evaluation of patients with neuromuscular disease and requirement of cough augmentation with MIE devices. The patients will undergo a randomised protocol of chest clearance with standard physio, low pressure and high pressure MIE. Data from this trial will allow an optimal treatment strategy to be developed and if data suggested would provide sufficient data to power an interventional trial to examine important clinical outcomes.

ELIGIBILITY:
Inclusion Criteria: STABLE

* Neuromuscular disease e.g. muscular dystrophy, motor neurons disease
* Respiratory muscle weakness (FVC <60%, snip <60%, sleep disordered breathing)
* Clinical evidence of respiratory secretions or cough PEF <270 and history of LRTI
* Documented clinical stability by supervising clinician

Inclusion Criteria: ACUTE

* Neuromuscular disease e.g. muscular dystrophy, motor neurons disease
* Respiratory muscle weakness (FVC <60%, snip <60%, sleep disordered breathing)
* Clinical evidence of respiratory secretions or cough PEF <270
* Admitted with respiratory deterioration

Exclusion Criteria: STABLE

* Decompensated respiratory failure (pH < 7.35)
* Pregnancy
* Aged <18, >80
* Change in ventilator settings in preceding 4 weeks
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Exclusion Criteria: ACUTE

* Decompensated respiratory failure (pH < 7.35), at time of recruitment
* Pregnancy
* Aged <18, >80
* Significant physical or psychiatric co-morbidity that would prevent compliance with trial protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction in the regional ventilation delays and Increase in homogeneity of ventilation post MIE vs baseline. | 1 day

SECONDARY OUTCOMES:
Change in neural respiratory drive (EMGpara) pre to post clearance | 1 day
  Change in neural respiratory drive (EMGpara) pre to post secretion clearance
Change in gas exchange (SpO2 and tcCO2) | 1 day
  Change in gas exchange, measured by taking SpO2 measurements and tCO2 measurements before and after secretion clearance
Subjective patient comfort (Visual analogue scale - VAS) | 1 day
  Change in patient comfort defined by VAS pre and post secretion clearance

CONTACTS AND LOCATIONS:
Locations (1):
- Guys and St Thomas NHS Foundation, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah NM, Apps C, Kaltsakas G, Madden-Scott S, Suh ES, D'Cruz RF, Arbane G, Patout M, Lhuillier E, Hart N, Murphy PB. The Effect of Pressure Changes During Mechanical Insufflation-Exsufflation on Respiratory and Airway Physiology. Chest. 2024 Apr;165(4):929-941. doi: 10.1016/j.chest.2023.10.015. Epub 2023 Oct 14. PMID 37844796